CLINICAL TRIAL: NCT00955760
Title: A Single Center, Open-Label, Three Periods, Fixed Sequence Design Study Analyzing the Effect of Rifampicin Administration on the Pharmacokinetics of Neramexane Mesylate
Brief Title: Study Analyzing the Effect of Rifampicin Administration on the Pharmacokinetics of Neramexane Mesylate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Michael Lissy, AAIPharma Deutschland GmbH & Co. KG
Masking: None
Other Study IDs: MRZ 92579/TI/1003
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — neramexane

INTERVENTIONS:
Drug: Neramexane — Drug-Drug Interaction Study

SUMMARY:
Primary Objectives:

• Assess the effects of poly-specific cytochrome P450 and drug-transporter induction by repeated dose Rifampicin (600 mg/day) co-administration on the single-dose pharmacokinetics of Neramexane.

Secondary Objectives:

• To assess safety and tolerability of Neramexane single dose treatment alone and co-administration of a Neramexane single dose with a Rifampicin repeated dose treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subject, who is able to read, to write and fully understand German language
* Aged 18 to 45 years (inclusive)
* BMI of 18-28 kg/m2 (inclusive) and a body weight of 50-90 kg (inclusive)
* Willing and able to provide written informed consent after having been informed of the requirements and the restrictions of the study
* Female subjects of childbearing potential must agree to use a highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1 % per year) when used consistently and correctly such as sexual abstinence, vasectomised partner, non hormonal IUDs, double barrier methods, e.g., condom and spermicide cream

Exclusion Criteria:

Safety concerns

* History of clinically relevant allergy or known hypersensitivity to Neramexane/Memantine/Amantadine and their derivatives
* History of clinically relevant allergy or known hypersensitivity to Rifampicin or other rifamycines
* History of clinically relevant allergy or known hypersensitivity to any inactive ingredient in any of the used investigational products or the metabolic inducer
* Exposure to another investigational agent within the last two months before Day 1 of Period 1
* Lactating or pregnant females or females planning to become pregnant during study conduct or within 2 months after end of study. Males planning to beget children during study conduct or within 2 months after end of study
* Any contraindications which are indicated in the topically valid SPC for EREMFAT®: severe hepatic impairment like obstructive jaundice, hepatitis, hepatic cirrhosis

Lack of suitability for the trial

* Any evidence of a significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, endocrinological, metabolic or other disease at screening
* History of malignancy
* Any clinically relevant deviation in clinical or laboratory assessment
* ECG abnormalities of clinical relevance, in particular abnormal prolongations of QT/QTc-interval (i.e., QTc ≥ 450 ms, PQ ≥ 220 ms)
* Systolic blood pressure < 95 mmHg or >150 mmHg or diastolic blood pressure < 50 mmHg or >90 mmHg in supine position
* Pulse rate <45 or >100 beats per minute
* Chronic or acute clinically relevant infections
* Chronic or acute disease, especially psychiatric or neurologic disorders
* History of alcohol or drug dependence
* Alcohol consumption averaging more than 40 g for male and more than 20 g for female subjects daily within the last year
* Regular caffeine consumption averaging more than 1 L of coffee and/or tea daily or more than 1 L of caffeine-containing lemonades per day within the last year
* Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal products (e.g., cholecystectomy, ulcus, etc.)
* Use of any prescribed medication for four weeks prior to the first administration of IMP.

  * Regular use of over-the-counter drugs [OTC] in the 4 weeks prior to the first administration of the IMP
  * Occasional use of OTC drugs (except paracetamol, maximum 1 g/day) within the 2 weeks prior to the first administration of the IMP.
  * Stable intake of thyroid hormone substitution will be allowed.
* Use of any food, food supplement or medication known to induce or inhibit CYP3A4 or other cytochrome P450 enzymes within two weeks preceding the start of the study (Day 1), e.g. grapefruit, St. John's wort
* Female subjects who employed any form of hormonal contraception within 2 months prior to study Day 1 (e.g. oral contraceptives, hormone releasing intrauterine contraceptive devices [IUDs], etc.)
* Consumption of xanthine derivates (including caffeine) within two days prior to Day 1
* Smoker and user of snuff, nicotine replacement and chewing tobacco
* Previous enrollment into the clinical phase of the current study
* Positive results in any of the serology tests
* Blood donation more than 450 mL within 60 days prior to Day 1
* Positive pregnancy test, if female
* Positive drug screen or alcohol test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AAIPharma Deutschland gmbH & Co. KG, Neu-Ulm, Bavaria, Germany